CLINICAL TRIAL: NCT05347914
Title: Mobile Mindfulness Intervention to Reduce Non-Homeostatic Food Cravings in Emotional Eaters: Research Pilot
Brief Title: Mindfulness App for Reducing Food Cravings
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McGill University (Other)
Responsible Party: Principal Investigator, Barbel Knauper, Professor, McGill University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: McGillU mindfulness app
Record Dates: First submitted 2022-04-16; First posted 2022-04-26 (Actual); Last update posted 2023-10-18 (Actual); Status verified 2023-10

CONDITIONS: Emotional Eating
MeSH Terms: conditions — Emotional Eating | interventions — Mindfulness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Mindfulness (Experimental)
  Interventions: Behavioral: Mindfulness

INTERVENTIONS:
Behavioral: Mindfulness — Participants will be taught a mindfulness exercise and will be instructed to use this exercise (following a mobile app) whenever they experience a food craving to eat for non-homeostatic reasons.

SUMMARY:
More than half of Canadian are overweight or obese and over fifty percent of individuals who are obese are emotional eaters. Emotional eating is defined as the tendency to eat in response to negative emotions and can be understood as reward-based eating behavior that is reinforced by modern obesogenic environments. Over time, food-related cues can interfere with reward-based learning processes such that an individual develops a conditioned response to eat for reasons that are not associated with physiological hunger. Mindfulness has the potential to act on the reward-base habit loop of emotional eating. One potential target is cravings or the urges to eat. This can be targeted using the mindfulness exercise called "RAIN" which calls for individuals to (1) Recognize and name their craving, to (2) Acknowledge its presence and to give it space to "be"; (3) then Investigate and bring an attitude of curiosity to their experience - Where did these feelings comes from? Have I felt this way before? then (4) Not-identify with your experience- that is, remind yourself that although your craving or urge to eat is very powerful, it only makes up a small part of who you are. The aim of the study is to therefore test a pilot intervention that implements a targeted mindfulness-based exercise (RAIN), using a mobile app, to attenuate the relationship between feeling a negative internal state (affect) and eating.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (age > 18 years) who meet criteria for emotional eating
2. Demonstrate a lack of control over eating
3. High levels of preoccupation with food

Exclusion Criteria:

1. Having been pregnant in the past six months or planning on becoming pregnant in the next year
2. currently undergoing treatment for cancer
3. using medication that affects body weight or appetite
4. being diagnosed with Bulimia Nervosa, Binge Eating Disorder, currently active Major Depression, or other psychiatric illnesses that may affect appetite.
5. Participants must also be proficient in English
6. Own a smartphone

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-08-28 (Actual); Study Completion 2023-08-28 (Actual)

PRIMARY OUTCOMES:
Change in food-related cravings | Baseline, week 6
  Food Craving Questionnaire Measures the frequency and intensity of food cravings in general. The 15-item scale assesses six dimensions of craving experiences: lack of control overeating, thoughts or preoccupation with food, intentions and plans to consume food, emotions before and during food cravings, as cues that may trigger food cravings. Items are rated on a scale of 1 (never) to 6 (always). Sample items include: "I feel like I have food on my mind all the time", "I crave foods when I feel bored, angry or sad" and "If I am craving something, thoughts of eating consume me". This measure has shown high internal consistency (Cronbach alphas between .80 and .91)
Change in emotional eating | Baseline, week 6
  Dutch Eating Behaviour Questionnaire The DEBQ is a 33-item self-report measure that assesses three dimensions of eating behaviours: emotion eating, restrained eating, and external eating. Individual are asked to indicate the extent to which they agree with each statement from 1 (seldom) to 5 (very often). Sample items include "Do you have a desire to eat when you are anxious, worried or tense?" and "If you see other eating, do you also have a desire to eat?". This measure has shown high internal consistency (Cronbach's alpha = .95)

SECONDARY OUTCOMES:
Change in feelings of control around eating | Baseline, week 6
  Brief Loss of Control Over-Eating Scale:
  The Brief Loss of Control Over-Eating Scale is a 7-item measure that assesses one's self-reported tendency to lose control over their eating behaviors. Items on the scale are rated from 1 (never) to 5 (always). Sample items include: "I felt like my cravings to eat overpowered me" and "I found myself eating despite negative consequences". The LOCES-B has shown high internal consistency (Cronbach alpha = .92)
Change in overidentification with food cravings | Baseline, week 6
  Cognitive Fusion Questionnaire- Food Cravings The Cognitive Fusion Questionnaire - Food Cravings is a (7-item) scale that assesses cognitive fusion with undesirable thoughts regards food craving and urges to eat. Sample items include: "It's very hard for me to let go of my food urges or cravings even when I know that letting go would be very helpful" and "I struggle to control my food urges or cravings." This measure has shown high internal consistency (Cronbach's alpha = .92).
Change in reactivity towards eating related experiences | Baseline, week 6
  UPPS-P Measure, Negative Urgency Scale:
  The UPPS-P Negative Urgency Scale is a 12-item measure that assess one's tendency to act rashly in response to negative mood states. Items on the scale are rated from 1 (I agree strongly) to 4 (I disagree strongly). Higher scores represent greater levels of impulsivity. Sample items include: "I have trouble controlling my impulses"). The UPPS-P Negative Urgency Scale has shown high internal consistency (Cronbach alpha = .88)
Change in judgment towards eating related experiences | Baseline, week 6
  Four Facet Mindful Eating Scale (FFaMES) The Four Facet Mindful Eating Scale is a 29-item self-report measure that assesses four dimensions of mindful eating: non-reactance, non-judgment, external awareness, and internal awareness. Individuals are asked to indicate the extent to which they agree with each statement from 1 (never) to 5 (very often). Sample items include: "I get carried away by my thoughts when I eat" and "I notice how the smell of food makes me want to eat." This measure has shown high internal consistency (non-reactance: Cronbach's alpha = .92, non-judgment: Cronbach's alpha = .91, external awareness: Cronbach's alpha = .82, internal awareness: Cronbach's alpha = .92).
Change in capacity to tolerate distress | Baseline, week 6
  Distress Tolerance Scale (DTS) The Distress Tolerance Scale is a 14-item scale that assesses an individual's ability to cope with various emotional states (e.g., happiness, anger, loneliness) that are in anticipating as well as in the present. Each item is rated on a scale of 1 (never) to 5 (all the time). Sample items include: "Felling distressed or upset is unbearable to me", "When I feel distressed or upset, all I can think about is how bad I feel" and "I can't handle feeling distressed or upset". The scale has shown high internal reliability (Cronbach's alpha = .91).

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - McGill University, Montreal, Please Select...
  - McGill University, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Anis AH, Zhang W, Bansback N, Guh DP, Amarsi Z, Birmingham CL. Obesity and overweight in Canada: an updated cost-of-illness study. Obes Rev. 2010 Jan;11(1):31-40. doi: 10.1111/j.1467-789X.2009.00579.x. Epub 2009 Apr 21. PMID 19413707
- [Background] Bongers P, de Graaff A, Jansen A. 'Emotional' does not even start to cover it: Generalization of overeating in emotional eaters. Appetite. 2016 Jan 1;96:611-616. doi: 10.1016/j.appet.2015.11.004. Epub 2015 Nov 10. PMID 26559754
- [Background] Born JM, Lemmens SG, Rutters F, Nieuwenhuizen AG, Formisano E, Goebel R, Westerterp-Plantenga MS. Acute stress and food-related reward activation in the brain during food choice during eating in the absence of hunger. Int J Obes (Lond). 2010 Jan;34(1):172-81. doi: 10.1038/ijo.2009.221. Epub 2009 Oct 20. PMID 19844211
- [Background] Brewer JA, Ruf A, Beccia AL, Essien GI, Finn LM, van Lutterveld R, Mason AE. Can Mindfulness Address Maladaptive Eating Behaviors? Why Traditional Diet Plans Fail and How New Mechanistic Insights May Lead to Novel Interventions. Front Psychol. 2018 Sep 10;9:1418. doi: 10.3389/fpsyg.2018.01418. eCollection 2018. PMID 30250438
- [Background] Cappelleri JC, Bushmakin AG, Gerber RA, Leidy NK, Sexton CC, Karlsson J, Lowe MR. Evaluating the Power of Food Scale in obese subjects and a general sample of individuals: development and measurement properties. Int J Obes (Lond). 2009 Aug;33(8):913-22. doi: 10.1038/ijo.2009.107. Epub 2009 Jun 9. PMID 19506564
- [Background] Carriere K, Shireen SH, Siemers N, Preissner CE, Starr J, Falk C, Knauper B. Development and Validation of the Four Facet Mindful Eating Scale (FFaMES). Appetite. 2022 Jan 1;168:105689. doi: 10.1016/j.appet.2021.105689. Epub 2021 Sep 10. PMID 34517074
- [Background] Dayan P, Niv Y. Reinforcement learning: the good, the bad and the ugly. Curr Opin Neurobiol. 2008 Apr;18(2):185-96. doi: 10.1016/j.conb.2008.08.003. Epub 2008 Aug 22. PMID 18708140
- [Background] Duarte C, Pinto-Gouveia J, Ferreira C, Silva B. Caught in the struggle with food craving: Development and validation of a new cognitive fusion measure. Appetite. 2016 Jun 1;101:146-55. doi: 10.1016/j.appet.2016.03.004. Epub 2016 Mar 2. PMID 26946280
- [Background] Elran Barak R, Shuval K, Li Q, Oetjen R, Drope J, Yaroch AL, Fennis BM, Harding M. Emotional Eating in Adults: The Role of Sociodemographics, Lifestyle Behaviors, and Self-Regulation-Findings from a U.S. National Study. Int J Environ Res Public Health. 2021 Feb 11;18(4):1744. doi: 10.3390/ijerph18041744. PMID 33670147
- [Background] Epel ES, Tomiyama AJ, Mason AE, Laraia BA, Hartman W, Ready K, Acree M, Adam TC, St Jeor S, Kessler D. The reward-based eating drive scale: a self-report index of reward-based eating. PLoS One. 2014 Jun 30;9(6):e101350. doi: 10.1371/journal.pone.0101350. eCollection 2014. PMID 24979216
- [Background] Epstein LH, Leddy JJ, Temple JL, Faith MS. Food reinforcement and eating: a multilevel analysis. Psychol Bull. 2007 Sep;133(5):884-906. doi: 10.1037/0033-2909.133.5.884. PMID 17723034
- [Background] Konttinen H, Mannisto S, Sarlio-Lahteenkorva S, Silventoinen K, Haukkala A. Emotional eating, depressive symptoms and self-reported food consumption. A population-based study. Appetite. 2010 Jun;54(3):473-9. doi: 10.1016/j.appet.2010.01.014. Epub 2010 Feb 4. PMID 20138944
- [Background] Latner JD, Mond JM, Kelly MC, Haynes SN, Hay PJ. The Loss of Control Over Eating Scale: development and psychometric evaluation. Int J Eat Disord. 2014 Sep;47(6):647-59. doi: 10.1002/eat.22296. Epub 2014 May 26. PMID 24862351
- [Background] Lee PC, Dixon JB. Food for Thought: Reward Mechanisms and Hedonic Overeating in Obesity. Curr Obes Rep. 2017 Dec;6(4):353-361. doi: 10.1007/s13679-017-0280-9. PMID 29052153
- [Background] Lowe MR, Butryn ML. Hedonic hunger: a new dimension of appetite? Physiol Behav. 2007 Jul 24;91(4):432-9. doi: 10.1016/j.physbeh.2007.04.006. Epub 2007 Apr 12. PMID 17531274
- [Background] Meule A, Teran CB, Berker J, Grundel T, Mayerhofer M, Platte P. On the differentiation between trait and state food craving: Half-year retest-reliability of the Food Cravings Questionnaire-Trait-reduced (FCQ-T-r) and the Food Cravings Questionnaire-State (FCQ-S). J Eat Disord. 2014 Sep 6;2(1):25. doi: 10.1186/s40337-014-0025-z. eCollection 2014. PMID 25356313
- [Background] Ozier AD, Kendrick OW, Leeper JD, Knol LL, Perko M, Burnham J. Overweight and obesity are associated with emotion- and stress-related eating as measured by the eating and appraisal due to emotions and stress questionnaire. J Am Diet Assoc. 2008 Jan;108(1):49-56. doi: 10.1016/j.jada.2007.10.011. PMID 18155989
- [Background] Papachristou H, Nederkoorn C, Beunen S, Jansen A. Dissection of appetitive conditioning. Does impulsivity play a role? Appetite. 2013 Oct;69:46-53. doi: 10.1016/j.appet.2013.05.011. Epub 2013 May 23. PMID 23707358
- [Background] Sinha R, Jastreboff AM. Stress as a common risk factor for obesity and addiction. Biol Psychiatry. 2013 May 1;73(9):827-35. doi: 10.1016/j.biopsych.2013.01.032. Epub 2013 Mar 26. PMID 23541000
- [Background] Sung J, Lee K, Song YM. Relationship of eating behavior to long-term weight change and body mass index: the Healthy Twin study. Eat Weight Disord. 2009 Jun-Sep;14(2-3):e98-105. doi: 10.1007/BF03327806. PMID 19934643
- [Background] Stice E, Burger K. Neural vulnerability factors for obesity. Clin Psychol Rev. 2019 Mar;68:38-53. doi: 10.1016/j.cpr.2018.12.002. Epub 2018 Dec 19. PMID 30587407
- [Background] Steward T, Menchon JM, Jimenez-Murcia S, Soriano-Mas C, Fernandez-Aranda F. Neural Network Alterations Across Eating Disorders: A Narrative Review of fMRI Studies. Curr Neuropharmacol. 2018;16(8):1150-1163. doi: 10.2174/1570159X15666171017111532. PMID 29046154
- [Background] Tomiyama AJ, Dallman MF, Epel ES. Comfort food is comforting to those most stressed: evidence of the chronic stress response network in high stress women. Psychoneuroendocrinology. 2011 Nov;36(10):1513-9. doi: 10.1016/j.psyneuen.2011.04.005. Epub 2011 Sep 8. PMID 21906885
- [Background] Van Gucht D, Baeyens F, Hermans D, Beckers T. The inertia of conditioned craving. Does context modulate the effect of counterconditioning? Appetite. 2013 Jun;65:51-7. doi: 10.1016/j.appet.2013.01.019. Epub 2013 Feb 10. PMID 23402718
- [Background] van Strien T, Herman CP, Verheijden MW. Eating style, overeating and weight gain. A prospective 2-year follow-up study in a representative Dutch sample. Appetite. 2012 Dec;59(3):782-9. doi: 10.1016/j.appet.2012.08.009. Epub 2012 Aug 20. PMID 22918175
- [Background] Ziauddeen H, Farooqi IS, Fletcher PC. Obesity and the brain: how convincing is the addiction model? Nat Rev Neurosci. 2012 Mar 14;13(4):279-86. doi: 10.1038/nrn3212. PMID 22414944